CLINICAL TRIAL: NCT04175470
Title: Bevacizumab and Tocotrienol in Recurrent Ovarian Cancer: A Marker Based Phase II Trial
Brief Title: Bevacizumab and Tocotrienol in Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BeTo-Ovar
Record Dates: First submitted 2019-11-14; First posted 2019-11-25 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — Bevacizumab; Tocotrienols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Discontinue treatment after first treatment cycle (Experimental)
  Interventions: Drug: Bevacizumab; Dietary Supplement: Tocotrienol
- Arm B: Continue treatment until progression (Experimental)
  Interventions: Drug: Bevacizumab; Dietary Supplement: Tocotrienol

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg intravenously every three weeks
Dietary Supplement: Tocotrienol — Capsules, 300 mg orally three times daily

SUMMARY:
A recent study at the Department of Oncology, Vejle Hospital (NCT02399592), investigated bevacizumab and tocotrienol in ovarian cancer patients and concurrently monitored the level of methylated HOXA9 circulating tumor DNA (HOXA9 meth-ctDNA) in the blood.

The rate of disease control was 70% with better results than other studies using bevacizumab alone. The toxicity was very low and attributed to bevacizumab only.

When the study results were worked up they showed that patients with a significant increase of HOXA9 meth-ctDNA after the first cycle of treatment did not benefit from the treatment whereas those with stable or decreasing HOXA9 meth-ctDNA did.

Therefore, in the current study patients with a high increase of HOXA9 meth-ctDNA after the first treatment cycle will discontinue treatment, as it is then considered ineffective. The remaining patients may achieve prolonged survival as predicted by their level of HOXA9 meth-ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian cancer, primary fallopian or primary peritoneal cancer.
* Platinum resistant epithelial ovarian cancer treated with at least two different previous chemotherapeutic regimens
* Progression on previous treatment. Previous treatment with bevacizumab is allowed.
* Measurable disease by the RECIST 1.1 criteria or evaluable by the GCIG CA-125 criteria.
* Age ≥ 18 years.
* Performance status 0-2.
* Adequate bone marrow function, liver function, and renal function (within 7 days prior to inclusion):

  * WBC ≥ 3.0 x 10^9/l or neutrophils (ANC) ≥ 1.5 x 10^9/l
  * Platelet count ≥ 100 x 10^9/l
  * Hemoglobin ≥ 6 mmol/l
  * Serum bilirubin < 2.0 x ULN
  * Serum transaminase ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 ULN
* Urine dipstick for protein < 2+. If the dipstick shows protein ≥ 2+, 24 hour urine testing must be performed and show protein contents < 1 g.
* Written informed consent

Exclusion Criteria:

* Other malignant disease within 3 years prior to inclusion in the study, except curatively treated basal cell or squamous cell carcinoma of the skin.
* Other experimental therapy or participation in another clinical trial within 28 days prior to treatment initiation.
* Intestinal infiltration or infiltration in major blood vessels at the discretion of the treating physician.
* Underlying medical disease not adequately treated (diabetes, cardiac disease).
* Uncontrolled hypertension (BP > 150/100 despite antihypertensive treatment).
* Surgery including open biopsy, within 4 weeks prior to first dose of bevacizumab.
* Cerebral vascular attack, transient ischemic attack or subarachnoid hemorrhage within 6 months before start of treatment.
* Clinical significant cardiovascular disease, including:

  * Myocardial infarction or unstable angina within 6 months before start of treatment
  * New York Heart Association (NYHA) class ≥ 2
  * Poorly controlled cardiac arrhythmia despite medication
  * Peripheral vascular disease grade ≥ 3
* Allergy to active substance or any of the auxiliary agents
* Bleeding tumor
* Pregnant or breast-feeding patients. For fertile women a negative pregnancy test at screening is mandatory.
* Fertile patients not willing to use effective methods of contraception during treatment and for 6 months after the end of treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 6 months after enrollment of the last patient

SECONDARY OUTCOMES:
Overall survival | 12 months after enrollment of the last patient
Response rate as measured by RECIST 1.1 or CA-125 | 6 months after enrollment of the last patient
Safety as measured by CTC version 5.0 | Every 9 weeks until progression, up to 3 years
  CTC = National Cancer Institute's Common Toxicity Criteria (NCI-CTC)

CONTACTS AND LOCATIONS:
Overall Officials: Torben F Hansen, MD, DMSc, Study Chair — Department of Oncology, Vejle Hospital - University Hospital of Southern Denmark
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark